CLINICAL TRIAL: NCT02724501
Title: Clinical and Molecular Studies of the Tumour Suppressor Gene PTEN in Endometrioid Type Endometrial Cancer
Brief Title: Studies of the Tumour Suppressor Gene PTEN - Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Trials Group (Network); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 01-0256-C; Terry Fox Grant #11425
Record Dates: First submitted 2011-02-11; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: questionnaire — Using questionnaire to obtain patient's medical and family history of cancer.
Procedure: Blood sample-DNA testing / Tumour-genetic markers — Using Samples obtained to produce summary statistics on the tumour markers

SUMMARY:
This project seeks to understand the role of the PTEN tumour suppressor gene in endometrial cancer (tumours of the uterine lining), the most common gynecologic cancer in the developed world. The studies in this program span the spectrum from fruit flies to humans, as part of a synergistic partnership that will significantly enhance our understanding of the molecular genetic events involved in the development and progression of endometrial cancer. The discovery of new targets for therapy, and the ability to evaluate these in subsequent clinical trials is a significant strength of this scientific interaction, which may result in cures for patients with primary and relapse endometrial cancer and prevention of this cancer in women who are at high risk.

DETAILED DESCRIPTION:
PTEN is a critical module that regulates effects of sex hormones on the growth and apoptosis of endometrial cells; and plays an important role in the pathogenesis of subgroups of endometrial cancers, their biologic behaviour and responses to therapeutic agents. Furthermore, mutational inactivation of the PTEN gene can serve as an independent molecular marker that can predict relapse and survival in endometrial cancer. The prognostic effects of PTEN may also be modulated by other tumour suppressor gene losses including P53 mutations, by hormone receptor status, and microsatellite instability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* patients who had a hysterectomy
* patient able to provide consent and complete questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Endometrial Cancer
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2000-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of endometrial cancer patients with inactivated PTEN tumor suppressor gene | 6 months
  Determining the association of PTEN inactivation and PKB expression, mutation of p53, microsatellite instability and progesterone receptor status in endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada